CLINICAL TRIAL: NCT01175330
Title: Randomized Trial of Fish Oil Infusion to Prevent Atrial Fibrillation After Cardiac Surgery
Brief Title: Omega 3 Fatty Acid Efficiency for Prevention of Atrial Fibrillation After Coronary Artery Bypass Grafting
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis did not reveal of anticipated benefits of intervention
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Efremov Sergey, Anesthesist, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAFPAF-042; MCAFS-042
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Ischemic Heart Disease; Atrial Fibrillation
Keywords: Omega-3 fatty acid; Ischemic Heart Disease; Atrial Fibrillation; Subcutaneous cardiac monitoring
MeSH Terms: conditions — Myocardial Ischemia; Atrial Fibrillation | interventions — fish oil triglycerides; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CABG and intralipid infusion (Placebo Comparator): Procedure: CABG surgery and subcutaneous cardiac monitor implantation Drug: Intralipid Lipid emulsion (Intralipid) for intravenous use, 1 ml/kg/day daily for 7 days post-surgery period (The first infusion beginning in operative period)
  Interventions: Drug: Intralipid
- CABG and omega-3 fatty acid infusion (Active Comparator): Procedure: CABG surgery and subcutaneous cardiac monitor implantation Drug: Omegaven Lipid emulsion (omegaven) for intravenous use, 1 ml/kg/day daily for 7 days post-surgery period (The first infusion beginning in operative period)
  Interventions: Drug: Omega-3 fish oil emulsion (Omegaven)

INTERVENTIONS:
Drug: Omega-3 fish oil emulsion (Omegaven) — Lipid emulsion (omegaven) for intravenous use, 1 ml/kg/day daily for 7 days post-surgery period (The first infusion beginning in operative period)
  Arms: CABG and omega-3 fatty acid infusion
Drug: Intralipid — Lipid emulsion (Intralipid) for intravenous use, 1 ml/kg/day daily for 7 days post-surgery period (The first infusion beginning in operative period)
  Arms: CABG and intralipid infusion

SUMMARY:
The purpose of this study is to evaluate efficacy of Polyunsaturated Fatty Acid for the prevention of Atrial Fibrillation and anti-inflammatory effects in patients after CABG surgery

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG surgery.
* Signed, documented informed consent prior to admission to the study.

Exclusion Criteria:

* Unstable angina, requiring intervention or CABG <24 hrs after screening.
* Decompensated congestive heart failure.
* Chronic, persistent, paroxysmal atrial fibrillation.
* Uncorrected significant valvular heart disease
* Known hypersensitivity to the study drug
* Left ventricular dysfunction (ejection fraction <35%)
* Use of anti-arrhythmic drugs other than beta blockers
* Non-cardiac illness with a life expectancy of less than 1 year
* Bleeding diathesis or history of coagulopathy
* Significant renal and liver insufficiency
* Significant thyroid, pulmonary disease
* Uncontrolled diabetes mellitus
* Patients on anti-arrhythmic drugs
* Patients with pacemaker
* Patients unable to provide/sign informed consent.
* Patients currently taking marine based omega-three fish oil supplements.
* Disturbances in lipid metabolism, serum triglyceride value >3 mmol/l

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Freedom of Atrial Fibrillation or other atrial arrhythmias | 2 years

SECONDARY OUTCOMES:
All cause mortality | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Patholody, Novosibirsk, Russia

REFERENCES:
- [Result] Lomivorotov VV, Efremov SM, Pokushalov EA, Romanov AB, Ponomarev DN, Cherniavsky AM, Shilova AN, Karaskov AM, Lomivorotov VN. Randomized trial of fish oil infusion to prevent atrial fibrillation after cardiac surgery: data from an implantable continuous cardiac monitor. J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1278-84. doi: 10.1053/j.jvca.2014.02.019. Epub 2014 Jul 11. PMID 25027101